CLINICAL TRIAL: NCT06601946
Title: Supporting Tools and Cognitive Aids for Lay Resuscitation - A Simulation Study
Brief Title: Supporting Tools and Cognitive Aids for BLS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christina Hafner, MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1346/2024
Record Dates: First submitted 2024-09-14; First posted 2024-09-19 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Basic Life Support (Simulation)

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- BLS Paper Based Cognitive Aid (Other)
  Interventions: Other: BLS Paper Based Cognitive App
- First Aid App (Other)
  Interventions: Other: First Aid App
- Corpatch App (Other)
  Interventions: Other: Corpatch App

INTERVENTIONS:
Other: BLS Paper Based Cognitive App — BLS Paper Based Cognitive App
  Arms: BLS Paper Based Cognitive Aid
Other: First Aid App — First Aid App
  Arms: First Aid App
Other: Corpatch App — Corpatch App
  Arms: Corpatch App

SUMMARY:
Various studies have shown that rapid and correctly performed cardiopulmonary resuscitation (CPR) significantly increases the survival rate after cardiac arrest. Such a situation can affect anyone, anywhere and at any time, making it all the more important to master the basic skills and abilities of Basic Life Support (BLS). Thanks to constant technical progress, there are now numerous digital tools in the field of lay resuscitation. There are also feedback devices for CPR for laypersons, the use of which is currently the subject of scientific debate. In order to evaluate the influence of various tools on the quality of lay resuscitation, we are planning a prospective, randomized study in a parallel group design. This study is aimed at medical laypersons between the ages of 18 and 70 who have completed a BLS course (e.g. first aid course for driver's license) within the last 10 years. All participants are asked to take part in a mannequin-based simulation scenario in a public place. As part of this simulation scenario, the BLS algorithm is to be performed (recognizing respiratory-circulatory arrest, calling for help, performing chest compressions, organizing a defibrillator). After performing the 1-minute cardiac massage, the scenario is ended. We plan to randomize into 3 groups. Group 1 will receive paper-based information material on how to perform BLS correctly. Group 2 will receive a first aid app. Group 3 will receive a small medical device (CorPatch®), which gives direct feedback on the quality of chest compressions (e.g. frequency, depth), including an accompanying app for support. The time to blood flow (defined as the succession of 5 sufficient chest compressions in this study) will be evaluated as the primary outcome. Secondarily, resuscitation management will be evaluated using a validated BLS checklist, the time to critical actions (such as time to alert the emergency services), the quality of CPR, the cognitive load of the participants and the user-friendliness of the assigned aid.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years
* First Aid Training within the last 10 years

Exclusion Criteria:

- medical student, physician, nurse, paramedic

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to blood flow | within 1 minute
  The time to blood flow (defined as the succession of 5 sufficient chest compressions in this study) will be evaluated as the primary outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria